CLINICAL TRIAL: NCT06742606
Title: Efficacy of Biological Therapy in Pediatric Inflammatory Bowel Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: biological therapy and IBD
Record Dates: First submitted 2024-11-22; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Effect of Drug
Keywords: biological therapy , IBD

STUDY DESIGN:
Intervention Model Description: patients diagnosed as IBD
  Inclusion Criteria:
  1. Age: patients diagnosed as IBD aged from 1 month to 16 years
  2. Patients fulfilling modified Porto criteria for diagnosis of IBD including clinical features, laboratory, radiological and pathological findings (Levine et al, 2014).
  3. Patients initially severely diseased or in relapse and planned to start or change biological therapy.
  Exclusion Criteria:
  1. Patients already on biological therapy and controlled.
  2. Patients with known humeral or cell mediated immunodeficiency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients diagnosed as IBD aged from 1 month to 16 years (Experimental): study will include 2 groups of pediatric IBD patients planned to start biological treatment or change to other biological therapy and each group formed of 20 patients Group
  1 of patients will receive Adalimumab while Group 1 will receive ustekinumab
  Interventions: Biological: Group 1 of patients will receive Adalimumab while Group 1 will receive ustekinumab

INTERVENTIONS:
Biological: Group 1 of patients will receive Adalimumab while Group 1 will receive ustekinumab — All the patients will be treated according to guidelines of ECCO/ESPGHAN and will be followed up regularly for 12 months by assessment
  • response to treatment Frequency of relapses,
  Regular assessment will be:
  Clinically every 2 to 4 weeks at gastroenterology outpatient clinic by using activity scoring systems:
  pediatric Ulcerative Colitis Activity Index pediatric Chron's Disease Activity Index
  Laboratory follow up will done at weeks 12,24,36,48 of starting or changing to other biological by doing inflammatory markers( CBC, ESR, CRP, albumin. At the end of study(week 48) each patient will be reassessed by:
  Disease activity:
  Laboratory Endoscopy will be repeated at week 48 of starting or changing to other biological to assess effect of biologicals on reach mucosal healing.

SUMMARY:
Compare efficacy of different biologicals in induction of remission including clinical, laboratory and histopathological remission.

DETAILED DESCRIPTION:
IBD are multifactorial disorders characterized by chronic relapsing intestinal inflammation (Fousekis et al .,2021). Main subtypes of pediatric IBD are Crohn's disease (CD), ulcerative colitis (UC), and IBD unclassified (Corica & Romano .., 2017) Mechanism of IBD involves uncontrolled immune mediated inflammatory response in genetically predisposed individuals to an unknown environmental trigger that interacts with gut microbiome and primarily affects gastrointestinal tract ( Iyer & Corr ..,2021) Pediatric onset IBD is more aggressive and rapidly progressive disease compared to adult onset IBD. Nearly a quarter of all patients with IBD develop this disease during childhood (Moon .., 2019), mean age at diagnosis ranged from 4.5 to 16 years in pediatric cases (Mosli et al ..,2021) Rates of pediatric onset IBD continue to rise around the world (Kuenzig et al ..,2022 ).

In2018, the highest annual incidences of pediatric IBD were 23/100000 person in Europe, 15.2/100000 in North America, and 11.4/100000 in Asia/ Middle East and Oceania (Sýkora et al .., 2018) Pediatric IBD management and therapeutic approach can be chall enging, especially in younger patients (Romeo et al .., 2020 )). Biologic agents have revolutionized the treatment paradigm of pediatric IBD (Kapoor & Crowley ..,2021) Biological drugs are monoclonal antibodies target specific cytokines involved in inflammatory cascade, such as tumour necrosis factor alpha (TNFα), integrins or interleukin 12/23, and have been approved for both pediatric CD and UC (Romeo et al 2020)

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling modified Porto criteria for diagnosis of IBD including clinical features, laboratory, radiological and pathological findings.

Patients initially severely diseased or in relapse and planned to start or change biological therapy.

Exclusion Criteria:

Patients already on biological therapy and controlled. Patients with known humeral or cell mediated immunodeficiency.

Ethical

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
Compare efficacy of different biologicals in induction of remission by histopathological remission using histological DCA scoring system | 48 weeks
  response to treatment Frequency of relapses, Control of symptoms and Following up growth pattern.
  histopathological scoring assessment will be by using Inflammatory Bowel Disease-Distribution, Chronicity, Activity [IBD-DCA] Score